CLINICAL TRIAL: NCT03392493
Title: The Effects on Hand Function With Robot-assisted Rehabilitation for Patients With Stroke
Brief Title: Robot-assisted Hand Rehabilitation for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB N201704068
Record Dates: First submitted 2017-08-24; First posted 2018-01-08 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Stroke; Robotic rehabilitation; Hand function; Activities of Daily Living
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: AB or BA
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): In the phase 1 :12 training sessions of Robot-assisted hand rehabilitation(60 minutes a time, 2 times a week); In the phase 2 :12 training sessions of Standard treatment only. (60 minutes a time, 2 times a week)
  Interventions: Behavioral: Robot-assisted hand rehabilitation; Behavioral: Standard treatment
- Group B (Active Comparator): In the phase 1 :12 training sessions of Standard treatment only(60 minutes a time, 2 times a week) ; In the phase 2 :12 training sessions of Robot-assisted hand rehabilitation(60 minutes a time, 2 times a week)
  Interventions: Behavioral: Robot-assisted hand rehabilitation; Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Robot-assisted hand rehabilitation — Robot-assisted hand rehabilitation: 20 minute of worm-up exercise and 40 minute of robot-assisted hand exercise. Robot-assisted hand exercises include passive range of motion of hand, bilateral hands task and robot-assisted task.
Behavioral: Standard treatment — Standard treatment only group: 60 min standard treatment. 20 minute of worm-up exercise and 40 minute of traditional occupational therapy. Traditional occupational therapy include spasticity-reducing activity, bilateral hands activity and hand training task.

SUMMARY:
Robotic therapy can deliver larger amounts of upper extremity movement practice for stroke rehabilitation. Although the treatment effects were supported in studies, there are still limitations in clinical intervention. The study will use the robot-assisted hand rehabilitation with a Gloreha device. Thirty patients with moderate motor deficits were recruited and randomized into 2 treatment groups, AB or BA (A = 12 times of robot-assisted hand rehabilitation, B = 12 times of standard therapy) for 12 weeks of treatment (Sixty minutes a time, twice a week), 1 month of break between conditions for washout period. The performance was assessed by a blinded assessor for five times (pre-test1, post-test 1, pre-test2, post-test 2, follow up at three month). The outcome measures Fugl-Meyer Assessment-Upper Limb section(FMA-UE),Box and block test(BBT), Maximal voluntary contraction(MVC) of extensor digitorum communis(EDC), Abductor pollicis brevis(APB), Flexor digitorum(FD), Dynanometer, Semmes-Weinstein hand monofilament (SWM), Revision of the Nottingham Sensory Assessment (EmNSA), Modified Barthel Index. Collected data will be analyzed with ANOVA test by SPSS version 20.0, and alpha level was set at 0.05. The hypothesis are robot-assisted hand rehabilitation with a Gloreha device has positive effects on sensory, motor, hand function, and ADL ability among patients with stroke.

DETAILED DESCRIPTION:
Many stroke survivors suffered problems with the upper extremity, such as paresis, synergy movement, hypertonicity, jag movement, sensory deficit. An inability to use the upper extremity in daily life can lead to loss of independence with ADLs and of important occupations (eg,work, driving). For individuals with more severe paresis, the potential for recovery of upper extremity function is greatly reduced. Robotic therapy can deliver larger amounts of upper extremity movement practice for these individuals. Although the Robotic therapy appears to provide some benefit for upper extremity motor abilities and participation but is of uncertain utility compared with dose-matched conventional upper limb exercise therapies. Objective: To investigate the effects of robot-assisted hand rehabilitation with a Gloreha device on sensory, motor, and ADL ability for patients with stroke.

Materials and Methods: Thirty patients with moderate motor deficits were recruited and randomized into 2 treatment groups, AB or BA (A = 12 times of robot-assisted hand rehabilitation, B = 12 times of standard therapy) for 12 weeks of treatment (Sixty minutes a time, twice a week), 1 month of break between conditions for washout period. The performance was assessed by a blinded assessor for five times (pre-test1, post-test 1, pre-test2, post-test 2, follow up at three month). The outcome measures Fugl-Meyer Assessment-Upper Limb section(FMA-UE),Box and block test(BBT), Maximal voluntary contraction(MVC) of extensor digitorum communis(EDC), Abductor pollicis brevis(APB), Flexor digitorum(FD), Dynanometer, Semmes-Weinstein hand monofilament (SWM), Revision of the Nottingham Sensory Assessment (EmNSA) for hand evaluations, Modified Barthel Index for ADL ability. Collected data will be analyzed with ANOVA test by SPSS version 20.0, and alpha level was set at 0.05. The hypothesis are robot-assisted hand rehabilitation with a Gloreha device has positive effects on sensory, motor, hand function, and ADL ability among patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* First stroke with hemiplegia
* Chronicity > 3 months
* Could understand the instructions
* Brunnstrom stageⅡ-Ⅴ
* Sensory impairment (Revision of the Nottingham Sensory Assessment-Tatile< 2; Kinaesthetic < 3)
* Modified Ashworth Scale < 3

Exclusion Criteria:

* Age younger than 20 and older than75 years
* Individuals with visual or auditory impairment who couldn't see or hear the feedback from the device clearly
* Individuals with other medical symptoms that can affect movement

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment：Upper Limb section | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Upper Limb motor function

SECONDARY OUTCOMES:
Box and block test | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Upper Limb motor function
EMG: record maximal voluntary contraction(MVC) of brachioradialis, extensor carpi, abductor pollicis longus | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Grip strength
Dynanometer | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Grip strength
Semmes-Weinstein hand monofilament | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Light touch
Revision of the Nottingham Sensory Assessment | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Proprioception
Modified barthel index | Change from baseline to 6 weeks, 10 weeks,16weeks, follow up at three month
  Activity of daily live ability

CONTACTS AND LOCATIONS:
Overall Officials: Jui chi Lin, master, Study Chair — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Department of Physical Medicine and Rehabilitation, Shuang Ho Hospital, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hatano S. Experience from a multicentre stroke register: a preliminary report. Bull World Health Organ. 1976;54(5):541-53. PMID 1088404
- [Background] Carod-Artal J, Egido JA, Gonzalez JL, Varela de Seijas E. Quality of life among stroke survivors evaluated 1 year after stroke: experience of a stroke unit. Stroke. 2000 Dec;31(12):2995-3000. doi: 10.1161/01.str.31.12.2995. PMID 11108762
- [Background] Chiu L, Shyu WC, Liu YH. Comparisons of the cost-effectiveness among hospital chronic care, nursing home placement, home nursing care and family care for severe stroke patients. J Adv Nurs. 2001 Feb;33(3):380-6. doi: 10.1046/j.1365-2648.2001.01703.x. PMID 11251725
- [Background] Nordin N, Xie SQ, Wunsche B. Assessment of movement quality in robot- assisted upper limb rehabilitation after stroke: a review. J Neuroeng Rehabil. 2014 Sep 12;11:137. doi: 10.1186/1743-0003-11-137. PMID 25217124
- [Background] Jang SH. The recovery of walking in stroke patients: a review. Int J Rehabil Res. 2010 Dec;33(4):285-9. doi: 10.1097/MRR.0b013e32833f0500. PMID 20805757
- [Background] Kopp B, Kunkel A, Muhlnickel W, Villringer K, Taub E, Flor H. Plasticity in the motor system related to therapy-induced improvement of movement after stroke. Neuroreport. 1999 Mar 17;10(4):807-10. doi: 10.1097/00001756-199903170-00026. PMID 10208552
- [Background] Basteris A, Nijenhuis SM, Stienen AH, Buurke JH, Prange GB, Amirabdollahian F. Training modalities in robot-mediated upper limb rehabilitation in stroke: a framework for classification based on a systematic review. J Neuroeng Rehabil. 2014 Jul 10;11:111. doi: 10.1186/1743-0003-11-111. PMID 25012864
- [Background] Correction to: Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e78. doi: 10.1161/STR.0000000000000120. No abstract available. PMID 28115727
- [Background] Susanto EA, Tong RK, Ockenfeld C, Ho NS. Efficacy of robot-assisted fingers training in chronic stroke survivors: a pilot randomized-controlled trial. J Neuroeng Rehabil. 2015 Apr 25;12:42. doi: 10.1186/s12984-015-0033-5. PMID 25906983
- [Background] Sivan M, O'Connor RJ, Makower S, Levesley M, Bhakta B. Systematic review of outcome measures used in the evaluation of robot-assisted upper limb exercise in stroke. J Rehabil Med. 2011 Feb;43(3):181-9. doi: 10.2340/16501977-0674. PMID 21305232
- [Background] Varalta V, Picelli A, Fonte C, Montemezzi G, La Marchina E, Smania N. Effects of contralesional robot-assisted hand training in patients with unilateral spatial neglect following stroke: a case series study. J Neuroeng Rehabil. 2014 Dec 5;11:160. doi: 10.1186/1743-0003-11-160. PMID 25476507
- [Background] Sgaggio, E., Joint and functional benefits of a robotic glove for post-stroke patients. publication pending, 2015.
- [Background] Pětioký, J. Robot-assisted therapy integrated with virtual reality for rehabilitation of hand function after stroke: a clinical case study. in the 20th ESPRM Congress 2016.
- [Background] Vanoglio F, Bernocchi P, Mule C, Garofali F, Mora C, Taveggia G, Scalvini S, Luisa A. Feasibility and efficacy of a robotic device for hand rehabilitation in hemiplegic stroke patients: a randomized pilot controlled study. Clin Rehabil. 2017 Mar;31(3):351-360. doi: 10.1177/0269215516642606. Epub 2016 Jul 10. PMID 27056250
- [Background] Mehrholz J, Hadrich A, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving generic activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD006876. doi: 10.1002/14651858.CD006876.pub3. PMID 22696362
- [Background] Cho KH, Lee KJ, Song CH. Virtual-reality balance training with a video-game system improves dynamic balance in chronic stroke patients. Tohoku J Exp Med. 2012 Sep;228(1):69-74. doi: 10.1620/tjem.228.69. PMID 22976384
- [Background] Zhang Y, Chapman AM, Plested M, Jackson D, Purroy F. The Incidence, Prevalence, and Mortality of Stroke in France, Germany, Italy, Spain, the UK, and the US: A Literature Review. Stroke Res Treat. 2012;2012:436125. doi: 10.1155/2012/436125. Epub 2012 Mar 1. PMID 22550614
- [Background] Ovbiagele B, Nguyen-Huynh MN. Stroke epidemiology: advancing our understanding of disease mechanism and therapy. Neurotherapeutics. 2011 Jul;8(3):319-29. doi: 10.1007/s13311-011-0053-1. PMID 21691873
- [Background] 民國100年衛生統計系列(一)死因統計及衛生統計系列(四)全民健康保險醫療統計. 2011: 行政院衛生署.
- [Background] O'Sullivan, S.B., T.J. Schmitz, and G. Fulk, Physical rehabilitation. 2013: FA Davis.
- [Background] Lang CE, Bland MD, Bailey RR, Schaefer SY, Birkenmeier RL. Assessment of upper extremity impairment, function, and activity after stroke: foundations for clinical decision making. J Hand Ther. 2013 Apr-Jun;26(2):104-14;quiz 115. doi: 10.1016/j.jht.2012.06.005. Epub 2012 Sep 10. PMID 22975740
- [Background] 黃琬倩, et al., 不同雙側上肢訓練模式對中風復健成效之文獻回顧. 職能治療學會雜誌, 2009. 27(第 2): p. P29-P48.
- [Background] Nilsen DM, Gillen G, Gordon AM. Use of mental practice to improve upper-limb recovery after stroke: a systematic review. Am J Occup Ther. 2010 Sep-Oct;64(5):695-708. doi: 10.5014/ajot.2010.09034. PMID 21073100
- [Background] Malouin F, Jackson PL, Richards CL. Towards the integration of mental practice in rehabilitation programs. A critical review. Front Hum Neurosci. 2013 Sep 19;7:576. doi: 10.3389/fnhum.2013.00576. PMID 24065903
- [Background] Wu CY, Huang PC, Chen YT, Lin KC, Yang HW. Effects of mirror therapy on motor and sensory recovery in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2013 Jun;94(6):1023-30. doi: 10.1016/j.apmr.2013.02.007. Epub 2013 Feb 15. PMID 23419791
- [Background] Lohse KR, Hilderman CG, Cheung KL, Tatla S, Van der Loos HF. Virtual reality therapy for adults post-stroke: a systematic review and meta-analysis exploring virtual environments and commercial games in therapy. PLoS One. 2014 Mar 28;9(3):e93318. doi: 10.1371/journal.pone.0093318. eCollection 2014. PMID 24681826
- [Background] Lohse K, Shirzad N, Verster A, Hodges N, Van der Loos HF. Video games and rehabilitation: using design principles to enhance engagement in physical therapy. J Neurol Phys Ther. 2013 Dec;37(4):166-75. doi: 10.1097/NPT.0000000000000017. PMID 24232363
- [Background] You SH, Jang SH, Kim YH, Hallett M, Ahn SH, Kwon YH, Kim JH, Lee MY. Virtual reality-induced cortical reorganization and associated locomotor recovery in chronic stroke: an experimenter-blind randomized study. Stroke. 2005 Jun;36(6):1166-71. doi: 10.1161/01.STR.0000162715.43417.91. Epub 2005 May 12. PMID 15890990
- [Background] Wuest S, van de Langenberg R, de Bruin ED. Design considerations for a theory-driven exergame-based rehabilitation program to improve walking of persons with stroke. Eur Rev Aging Phys Act. 2014;11(2):119-129. doi: 10.1007/s11556-013-0136-6. Epub 2013 Dec 7. PMID 25309631
- [Background] Vernadakis N, Derri V, Tsitskari E, Antoniou P. The effect of Xbox Kinect intervention on balance ability for previously injured young competitive male athletes: a preliminary study. Phys Ther Sport. 2014 Aug;15(3):148-55. doi: 10.1016/j.ptsp.2013.08.004. Epub 2013 Sep 4. PMID 24239167
- [Background] Pichierri G, Wolf P, Murer K, de Bruin ED. Cognitive and cognitive-motor interventions affecting physical functioning: a systematic review. BMC Geriatr. 2011 Jun 8;11:29. doi: 10.1186/1471-2318-11-29. PMID 21651800
- [Background] Peters DM, McPherson AK, Fletcher B, McClenaghan BA, Fritz SL. Counting repetitions: an observational study of video game play in people with chronic poststroke hemiparesis. J Neurol Phys Ther. 2013 Sep;37(3):105-11. doi: 10.1097/NPT.0b013e31829ee9bc. PMID 23872681
- [Background] Rong W, Tong KY, Hu XL, Ho SK. Effects of electromyography-driven robot-aided hand training with neuromuscular electrical stimulation on hand control performance after chronic stroke. Disabil Rehabil Assist Technol. 2015 Mar;10(2):149-59. doi: 10.3109/17483107.2013.873491. Epub 2013 Dec 31. PMID 24377757
- [Background] Yun GJ, Chun MH, Park JY, Kim BR. The synergic effects of mirror therapy and neuromuscular electrical stimulation for hand function in stroke patients. Ann Rehabil Med. 2011 Jun;35(3):316-21. doi: 10.5535/arm.2011.35.3.316. Epub 2011 Jun 30. PMID 22506139
- [Background] Sharma, P., J.M. Sutaria, and P. Zambare, Effects of Neuromuscular Electrical Stimulation (NMES) on Hand Function in Stroke Patients. Indian Journal of Physiotherapy and Occupational Therapy-An International Journal, 2015. 9(3): p. 43-48.
- [Background] Carey, L.M., Somatosensory loss after stroke. Critical Reviews™ in Physical and Rehabilitation Medicine, 1995. 7(1).
- [Background] Pumpa LU, Cahill LS, Carey LM. Somatosensory assessment and treatment after stroke: An evidence-practice gap. Aust Occup Ther J. 2015 Apr;62(2):93-104. doi: 10.1111/1440-1630.12170. Epub 2015 Jan 23. PMID 25615889
- [Background] Carey LM, Matyas TA, Oke LE. Sensory loss in stroke patients: effective training of tactile and proprioceptive discrimination. Arch Phys Med Rehabil. 1993 Jun;74(6):602-11. doi: 10.1016/0003-9993(93)90158-7. PMID 8503750
- [Background] Smania N, Montagnana B, Faccioli S, Fiaschi A, Aglioti SM. Rehabilitation of somatic sensation and related deficit of motor control in patients with pure sensory stroke. Arch Phys Med Rehabil. 2003 Nov;84(11):1692-702. doi: 10.1053/s0003-9993(03)00277-6. PMID 14639572
- [Background] Dobkin BH. Strategies for stroke rehabilitation. Lancet Neurol. 2004 Sep;3(9):528-36. doi: 10.1016/S1474-4422(04)00851-8. PMID 15324721
- [Background] Buerger, S.P. and N. Hogan. Relaxing passivity for human-robot interaction. in 2006 IEEE/RSJ International Conference on Intelligent Robots and Systems. 2006. IEEE.
- [Background] Volpe BT, Lynch D, Rykman-Berland A, Ferraro M, Galgano M, Hogan N, Krebs HI. Intensive sensorimotor arm training mediated by therapist or robot improves hemiparesis in patients with chronic stroke. Neurorehabil Neural Repair. 2008 May-Jun;22(3):305-10. doi: 10.1177/1545968307311102. Epub 2008 Jan 9. PMID 18184932
- [Background] Hasegawa Y, M.Y., Watanabe K, Sankai Y, Five-fingered assistive hand with mechanical compliance of human finger. In IEEE Int. Conf.Robotics and Automation (ICRA). Pasadena, CA, 2008: p. 718-724.
- [Background] Rocon E, Belda-Lois JM, Ruiz AF, Manto M, Moreno JC, Pons JL. Design and validation of a rehabilitation robotic exoskeleton for tremor assessment and suppression. IEEE Trans Neural Syst Rehabil Eng. 2007 Sep;15(3):367-78. doi: 10.1109/TNSRE.2007.903917. PMID 17894269
- [Background] Loureiro RCV, B.-L.J., Lima ER, Pons JL, Sanchez-Lacuesta JJ,Harwin WS, Upper limb tremor suppression in ADL via an orthosis incorporating a controllable double viscous beam actuator. In Proc. 9th Int. Conf. on Rehabilitation Robotics ICORR. Chicago, IL, 2005: p. 119-122.
- [Background] Pedrocchi A, Ferrante S, Ambrosini E, Gandolla M, Casellato C, Schauer T, Klauer C, Pascual J, Vidaurre C, Gfohler M, Reichenfelser W, Karner J, Micera S, Crema A, Molteni F, Rossini M, Palumbo G, Guanziroli E, Jedlitschka A, Hack M, Bulgheroni M, d'Amico E, Schenk P, Zwicker S, Duschau-Wicke A, Miseikis J, Graber L, Ferrigno G. MUNDUS project: MUltimodal neuroprosthesis for daily upper limb support. J Neuroeng Rehabil. 2013 Jul 3;10:66. doi: 10.1186/1743-0003-10-66. PMID 23822118
- [Background] Chang WH, Kim YH. Robot-assisted Therapy in Stroke Rehabilitation. J Stroke. 2013 Sep;15(3):174-81. doi: 10.5853/jos.2013.15.3.174. Epub 2013 Sep 27. PMID 24396811
- [Background] Dijkers MP, deBear PC, Erlandson RF, Kristy K, Geer DM, Nichols A. Patient and staff acceptance of robotic technology in occupational therapy: a pilot study. J Rehabil Res Dev. 1991 Spring;28(2):33-44. doi: 10.1682/jrrd.1991.04.0033. PMID 2066869
- [Background] Fasoli SE, Krebs HI, Ferraro M, Hogan N, Volpe BT. Does shorter rehabilitation limit potential recovery poststroke? Neurorehabil Neural Repair. 2004 Jun;18(2):88-94. doi: 10.1177/0888439004267434. PMID 15228804
- [Background] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Background] Hsieh YW, Wu CY, Lin KC, Yao G, Wu KY, Chang YJ. Dose-response relationship of robot-assisted stroke motor rehabilitation: the impact of initial motor status. Stroke. 2012 Oct;43(10):2729-34. doi: 10.1161/STROKEAHA.112.658807. Epub 2012 Aug 14. PMID 22895994
- [Background] Lincoln, N., J. Jackson, and S. Adams, Reliability and revision of the Nottingham Sensory Assessment for stroke patients. Physiotherapy, 1998. 84(8): p. 358-365.
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Background] Bell-Krotoski J, Tomancik E. The repeatability of testing with Semmes-Weinstein monofilaments. J Hand Surg Am. 1987 Jan;12(1):155-61. doi: 10.1016/s0363-5023(87)80189-2. PMID 3805636